CLINICAL TRIAL: NCT04609891
Title: A Single-arm, Multi-center, Open Clinical Study of Avatrombopag on the Treatment of Thrombocytopenia Induced by Chemotherapy of Malignant Tumors
Brief Title: Avatrombopag on the Treatment of Thrombocytopenia Induced by Chemotherapy of Malignant Tumors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Anhui Provincial Cancer Hospital (Other)
Responsible Party: Principal Investigator, Qian Liting, Professor, Anhui Provincial Cancer Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SKXCIT001
Record Dates: First submitted 2020-10-04; First posted 2020-10-30 (Actual); Last update posted 2022-04-29 (Actual); Status verified 2022-04

CONDITIONS: Thrombocytopenia
Keywords: chemotherapy; rh-TPO; avatrombopag
MeSH Terms: conditions — Thrombocytopenia | interventions — avatrombopag

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Avatrombopag Tablets Oral (Experimental): When patient is diagnosed with thrombocytopenia induced by chemotherapy of malignant tumor, avatrombopag will be given to patients as a therapeutic plan.
  Interventions: Drug: Avatrombopag

INTERVENTIONS:
Drug: Avatrombopag — 10×109/L<PLT<75×109/L, avatrombopag tablet 60 mg once a day for 5-10 days.

SUMMARY:
To observe the clinical efficacy and safety of avatrombopag for chemotherapy-induced thrombocytopenia in patients with malignant tumors.

DETAILED DESCRIPTION:
Tumor is one of the malignant diseases that people face. In 2015, the incidence of malignant tumors was about 3.929 million, and the annual growth rate is about 3.9%. Chemotherapy is currently the most commonly used treatment for patients with tumor, but chemotherapy also brings many other problems, such as thrombocytopenia which can leads to increased medical costs, chemotherapy cycles delayed, and chemotherapy doses reduced. Studies have found that the reduction of the chemotherapy dose and the delay of the chemotherapy cycle will affect the survival rate of patients. So it is an important to solve the problem of chemotherapy-induced thrombocytopenia.

Currently, there are some methods to treat thrombocytopenia such as platelet transfusion, rhTPO, rhIL-11 and other methods. However, these methods have some defects, platelets are at risk of ineffective transfusion, rhTPO may produce neutralizing antibodies and rhIL-11 has serious side effects. Therefore, there is an urgent need for safer and faster methods to treat chemotherapy-induced thrombocytopenia. As a new generation of TPO receptor agonist, avatrombopag has the advantages of being taken with food, no hepatotoxicity, good safety, and rapidly increase platelet count. Therefore, avatrombopag has great research value in the treatment of chemotherapy-induced thrombocytopenia.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, aged 18~75 years.
2. Diagnosed with malignant tumors (gynecological tumors, gastrointestinal tumors, lung cancer, gastric cancer and head and neck tumors) by pathology or cytology and need chemotherapy.
3. The subject had developed at least grade II thrombocytopenia after the last chemotherapy cycle (10×109/L<PLT count<75×109/L).
4. Subjects' Eastern Cooperative Oncology Group (ECOG) performance status score ≤ 2.
5. The subjects' life expectancy at the time of screening is ≥12 weeks, and must continue to receive at least 2 cycles of the same chemotherapy regimen at the time of screening.
6. Women of childbearing age must have taken reliable contraceptive measures, or have a pregnancy test (serum or urine) within 7 days before enrollment, and the result is negative, and are willing to use appropriate methods of contraception during the trial.
7. The subjects voluntarily and strictly abide by the requirements of the research protocol and sign a written informed consent.

Exclusion Criteria:

1. Subjects suffer from severe cardiovascular disease: myocardial ischemia or myocardial infarction above grade II, poorly controlled arrhythmia; according to NYHA standards, grade III to IV cardiac insufficiency, or cardiac color Doppler ultrasound examination suggests left ventricular ejection fraction ( LVEF) <50%.
2. Subjects have clinically significant acute or active bleeding (such as gastrointestinal or central nervous system) within 7 days before screening.
3. Subjects received major surgery or minor surgery within 4 weeks of enrollment ≤ 3 days.
4. Subjects had a history of arterial or venous thrombosis (such as myocardial ischemia, transient ischemic attack, or stroke) within 6 months before screening.
5. Subjects had active infection or acute infection occurred within 2 weeks before the first administration of the study.
6. Long-term bed rest, subjects with severe vascular disease.
7. Subjects had a history of chronic thrombocytopenia or bleeding disorders, or a history of thrombocytopenia (such as chronic liver disease or immune thrombocytopenic purpura) caused by causes other than thrombocytopenia caused by chemotherapy.
8. Subjects had a history of other malignant tumors, such as acute lymphoblastic leukemia, acute myeloid leukemia, any myeloid malignant tumor, myelodysplastic syndrome, myeloproliferative disease, and multiple myeloma.
9. There are factors that significantly affect the absorption of oral drugs, such as inability to swallow, chronic diarrhea, and intestinal obstruction.
10. Subjects had an allergic reaction to avatrombopag or any of its excipients.
11. Subjects participated in clinical studies of other study drugs or devices within 30 days before screening.
12. The investigator assessed that the subjects had any accompanying medical history that could impair the subject's safety in completing the study, such as renal failure due to hemodialysis or active infection requiring intravenous antibiotics.
13. Subjects had a history of psychotropic drug abuse and unable to quit or have mental disorders.
14. Pregnant or breastfeeding women, and fertile patients who are unwilling or unable to take effective contraceptive measures.
15. The investigator judges other conditions that may affect the conduct of clinical research and the determination of research results.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2020-05-26 (Actual); Primary Completion 2021-05-16 (Actual); Study Completion 2021-05-16 (Actual)

PRIMARY OUTCOMES:
Proportion of responders | up to 2 months
  Proportion of patients with platelet count ≥100×10^9/L or increase of platelet count ≥50×10^9/L or ≥100% from baseline within cycle X after initiation of avatrombopag treatment.Due to chemotherapy induced thrombocytopenia in the X+1 cycle, the dose reduction in chemotherapy of X+2 cycle by ≥15% or chemotherapy delay by ≥4 days.

SECONDARY OUTCOMES:
Duration of grade Ⅲ and Ⅳ thrombocytopenia after initiation of avatrombopag treatment | up to 2 months
Time for PLT to recover to ≥75×10^9/L and ≥100×10^9/L after initiation of avatrombopag treatment | up to 2 months
minimal platelet count | up to 2 months
Proportion of patients without platelet transfusion | up to 2 months
Proportion of patients without bleeding | up to 2 months

CONTACTS AND LOCATIONS:
Locations (1):
- Anhui Provincial Cancer Hospital, Hefei, Anhui, China

REFERENCES:
- [Derived] Cui Y, He Y, Hu C, Tu C, Huang J, Zhu X, Zang C, Ding K, Zhan B, Zhao Y, Qian L. Avatrombopag for the treatment of thrombocytopenia induced by chemotherapy in patients with solid tumors: A multicenter, open-label, single-arm trial. Front Pharmacol. 2022 Sep 27;13:970978. doi: 10.3389/fphar.2022.970978. eCollection 2022. PMID 36238568